CLINICAL TRIAL: NCT05259514
Title: The Efficacy of CytoSorb in the Removal of IL-6 in Severe Aneurysmal Subarachnoid Hemorrhage - a Two Phase Study - a Primary Feasibility Study (Phase 1) - a Secondary Randomized, Controlled, Prospective Proof-of-concept Study (Phase 2)
Brief Title: CytoSorb SAH Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: safety
Sponsor: Emanuela Keller (Other)
Collaborators: CytoSorbents Europe GmbH (Industry)
Responsible Party: Sponsor-Investigator, Emanuela Keller, Prof. Dr., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-D0082
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Aneurysmal Subarachnoid Haemorrhage

STUDY DESIGN:
Intervention Model Description: study phase 1 (feasibility/power-analysis): 5 treated with CytoSorb study phase 2: 40 (20 standard of care and 20 Cytosorb).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CytoSorb (Experimental): Phase 2: 40 (20 each in treatment and control group). The Study Product is CytoSorb. Patients included will receive a CytoSorb filter. The device has a CE-mark and is used in accordance with its CE-Certification. Patients are installed as early as possible after exclusion of the bleeding source and are treated with the CytoSorb Adsorber for 48 hours. Blood flow will be set at least 200 ml/min.
  Interventions: Device: CytoSorb
- Standard of Care (No Intervention): Only routine treatment

INTERVENTIONS:
Device: CytoSorb — The Study Product is CytoSorb. Patients included will receive a CytoSorb filter. The device has a CE-mark and is used in accordance with its CE-Certification. Patients are installed as early as possible after exclusion of the bleeding source and are treated with the CytoSorb Adsorber for 48 hours. Blood flow will be set at least 200 ml/min.
  Arms: CytoSorb

SUMMARY:
In aSAH high levels of IL-6 (a pro-inflammatory cytokine) in the cerebrospinal fluid, as well as systemically have been linked to the severity grade and the occurrence of vasospasm and delayed cerebral ischemia caused by vasospasm as well as worse outcome independent of severity grade at time of admission and age. Increased levels of IL-6 increase the probability of unfavourable outcome, as well as the occurrence of delayed ischemic neurological deficit.

CytoSorb is an available, and certified medical device intended for use in conditions where elevated levels of cytokines such as IL-6 exist. Its clinical effect lies in the reduction of levels of pro-inflammatory mediators and thereby improving organ function as well as improving hemodynamic stability within hours of treatment initiation. Currently it is primarily used for the treatment of patients with confirmed or imminent respiratory failure who have either an acute lung injury, or acute respiratory distress syndrome, or a severe disease incl. respiratory failure, septic shock, and or multiple organ dysfunction/failure.

Until now, effective IL-6 removal in patients suffering from aSAH has not been possible in human and thus has not yet been evaluated. The purpose of this study is to see whether removal of IL-6 in patients with aSAH using CytoSorb is possible, and whether this alters the clinical course.

The overall goal of this study is to investigate whether a treatment with CytoSorb removes Interleukin 6 in patients with aSAH, and whether the treatment with CytoSorb alters the clinical course.

DETAILED DESCRIPTION:
Study phase 1: patients (not randomized) will be allocated to the treatment group and compared to an already existing retrospective control group. The measurements and procedures are otherwise the same as in phase 2: Patients are randomized into a treatment group and a control group. In the treatment group the study intervention consists of the installation of a central venous line, connected to a device for hemoperfusion and removal of IL-6 using a CytoSorb Adsorber.

The overall objective is to evaluate efficacy, IL-6 levels will be measured daily in blood plasma as well as in cerebrospinal fluid between day 1 up to day 14 (routine procedure). Plasma and cerebrospinal fluid levels of IL-6 are evaluated using the routine samples. Furthermore, IL-6 will also be measured right after Cytosorb and the filtration to evaluate the amount of IL-6 that is actually removed by the filter (study-specific).

Only post-filter blood samples are taken for study purposes. Two post-filter blood samples (10-20ml totally) are taken for study purposes: first sample one hour after installation of CytoSorb and the second sample: 24 hours after installation.

Patient in the control group have standard of care treatment. The usual standard of care for the management of aneurysmal subarachnoid haemorrhage will be performed during the entire treatment period in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age ≥ 18years) admitted to the Neurointensive Care Unit (NICU)
* Subjects with aSAH with external ventricular drainage on admission computed tomography (CT) scan due to a ruptured aneurysm confirmed by digital subtracted angiography (DSA) or computed tomography based angiography (CTA), and successfully secured aneurysm by clipping or coiling within 3 days after aneurysm rupture
* Admission WFNS grade 4-5 (high-grade aSAH)
* A physician who is not participating in the research project is called in to safeguard the interests of the person concerned before he or she is involved in the project
* Informed Consent by signature from representative
* Informed Consent (post-hoc) by signature from patient, if possible

Exclusion Criteria:

* Subjects with moderate to severe vasospasm at time of admission as confirmed by CTA or DSA
* Any severe or unstable known inflammatory/immunodeficiency condition or disease (e.g. cancer, haematological, chronic infection or autoimmune disease) that might alter the natural inflammatory response
* Patients concurrently requiring immunosuppressive therapy, or who are profoundly immune suppressed
* Current infection with necessity of antibiotic treatment
* Any known coagulopathy or history of thromboembolic event leading to increased risk for thrombosis or bleeding
* Known allergies to polystyrene/divinylbenzene, polycarbonate, polypropylene, silicone and polyester
* Current pregnancy (as evaluated using a pregnancy test)
* Patients with very low platelet counts (< 20,000/μL).
* History of heparin-induced thrombocytopenia
* Acute sickle cell crisis
* Morbid obesity with BMI ≥ 40 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Reduction of plasma level of Interleukin-6 in patients with aSAH. | 14 days
  The primary objective is to determine, whether CytoSorb effectively reduces the plasma levels of Interleukin (IL)-6 in patients with aSAH.

SECONDARY OUTCOMES:
Reduction of IL-6 level within CSF | 14 days
  To evaluate whether CytoSorb effectively reduces the level of IL-6 within cerebrospinal fluid
Removal of IL-6 | 14 days
  To evaluate the amount of IL-6 that is removed

OTHER OUTCOMES:
Frequency of occurrence of aSAH specific complications | 14 days
  To evaluate whether CytoSorb alters the frequency of occurrence of aSAH specific complications in (as vasospasm/DCI) in comparison to the control group as well as the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland